CLINICAL TRIAL: NCT00530257
Title: Effect of OROS-Methylphenidate (Concerta) on Different Domains of Attention and Working Memory in Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: Study of the Effects of Osmotic-Release Oral System (OROS) Methylphenidate (Concerta) on Attention and Memory
Acronym: CHOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004-3-3588
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Methylphenidate; Attention; Working Memory
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (sugar pill);Subjects will be equally randomized and will receive one week of treatment with placebo and compared to subjects who were randomized to receive one week of OROS-methylphenidate.
  Interventions: Drug: Placebo
- OROS-methylphenidate (Active Comparator): Subjects will be equally randomized and will receive one week of treatment with the optimal dose of OROS methylphenidate compared with subjects randomized to receive one week of placebo.
  Interventions: Drug: OROS-methylphenidate

INTERVENTIONS:
Drug: Placebo — Placebo (sugar pill)
  Arms: Placebo
Drug: OROS-methylphenidate — 18 mg to 54 mg once a day for 1 week
  Other Names: Concerta; Osmotic-Release Oral System -methylphenidate
  Arms: OROS-methylphenidate

SUMMARY:
This study investigates whether OROS-methylphenidate improves performance on different aspects of attention and memory in children with Attention-Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
This study investigates the effect of Osmotic-Release Oral System (OROS)-methylphenidate, a long-acting stimulant, on multiple dimensions of attention and on working memory. Specifically, we will investigate the following two hypotheses: (1) OROS-methylphenidate will result in improved performance on measures assessing multiple domains of attention, including sustained attention, attentional control, selective attention, and divided attention, and (2) OROS-methylphenidate will result in improved performance on measures of working memory. In addition we will use the study to collect pilot data on whether the magnitude of the effect of OROS-methylphenidate varies across the different components of attention and working memory and whether improvement across any of these measures is helpful in predicting parent or teacher ratings of improvement.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual-IV Edition (DSM-IV) Criteria for ADHD.Combined Type
* Parent and Teacher Ratings >85 percentile on inattention and/or hyperactivity/impulsivity scales
* Estimated Intelligence Quotient (IQ) > 80 on Wechsler Abbreviated Scale of Intelligence or similar IQ test

Exclusion Criteria:

* Past or current diagnosis of Tourette syndrome or chronic tic disorder, Pervasive Developmental Disorder (PDD), Cerebral Palsy, Head Injury requiring hospitalization, psychotic disorder, hypertension, glaucoma, cardiovascular disease, severe narrowing of the gastrointestinal tract, or epilepsy
* Current diagnosis of bipolar disorder, obsessive-compulsive disorder serious enough to warrant separate treatment, suicidal or homicidal behavior or ideation
* Use within 14-days of a monoamine oxidase inhibitor
* History of side effects on any methylphenidate preparation that required stopping the medication
* Inability to swallow a capsule or tablet
* Chronic treatment with coumarin, clonidine, or tricyclic antidepressants

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2004-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan J Blum, M.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from an outpatient ADHD evaluation and treatment program at a pediatric academic medical center. Eligible children wer: 1) Age 6-12 years and at least in 1st grade; 2) DSM-IVTR diagnosis of ADHD, Combined Type;3) Parent and teacher ratings on the ADHD Rating Scale-IV > 85th percentile; 5) IQ greater than 75
Pre-assignment Details: Parents of 41 patients inquired about participating in the study. Four did not meet eligibility requirements leaving 37 eligible children. Three families elected not to participate leaving 34 children. Three children did not complete the dose finding stage leaving 31 children who entered the double blind placebo controlled crossover study.
Groups:
- OROS Methylphenidate: Children participated in a double blind placebo controlled crossover study comparing one week of treatment with the optimal dose of OROS methylphenidate with one week of treatment with placebo. The order of administering OROS-methylphenidate versus placebo was randomized and counterbalanced across participants. At the end of each week the child's performance on different domains of attention and executive functioning was assessed on the measures described below.
Period: Overall Study
Arm/Group | OROS Methylphenidate
Started | 31
Completed | 30
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | OROS Methylphenidate
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.5 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Test of Everyday Attention for Children: Walk, Don't Walk
Description: The TEA-Ch is a battery of nine subtests designed to assess multiple attentional capacities in children 6-16y.o. The Walk-Don't Walk subtest is a measure of sustained attention and response inhibition. Scores on this subtest can range from 0 to 20 with higher scores representing better performance.
Time Frame: 2 weeks
Population: Crossover design, all 30 of the 31 subjects completed both the placebo and medication phase of the study and were the group analyzed
Measure: Median (Full Range); unit: units on a scale
Groups:
- Medication: Children participated in a double blind placebo controlled crossover study comparing one week of treatment with the optimal dose of OROS methylphenidate with one week of treatment with placebo. The order of administering OROS-methylphenidate versus placebo was randomized and counterbalanced across participants. At the end of each week the child's performance on different domains of attention and executive functioning was assessed.
- Placebo: This is a crossover study. Thirty of thirty-one enrolled subjects completed the medication and placebo phases
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 13.5 [0 to 20] | 11 [0 to 19]
Statistical Analysis 1: Comparison: Medication vs Placebo; We evaluated the data for cross over effects. No statistical significant sequence effect were seen for our endpoints and hence we combined the data from both periods of the crossover design There was evidence against the assumption of normality for performance on some of the measures of attention. Thus we used the non-parametric Wilcoxon Signed Ranks Test to compare performance on OROS-methylphenidate versus placebo; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney) — We used a Bonferroni correct to adjust for up to 5 measures across domains and use a p-value of <=0.01. With a sample of 30 subjects the analytic model was able to detect a difference of large effect size (Cohen's d= >0.655)

2. Primary Outcome: Gordon Diagnostic System Continuous Performance Test
Description: This is a measure of sustained attention & response inhibition for children 6 yrs and older. During this task a series of numbers flash, one at a time, on a screen. The subject is told to press a button every time a "1" is followed by a "9". There are 45 possible correct responses over the 9-minute task. Omission errors are a measure of sustained attention and can range from 0 to 45. Commission errors are a measure of sustained attention and response inhibition can range from zero to hundreds (each time the button is pushed at the incorrect time). Lower scores indicate better performance.
Time Frame: 2 weeks
Population: 31 participants began the crossover phase of the trial and 30 completed both the medication and placebo arms. For one patient there was an equipment problem so that subject did not have data available
Measure: Median (Full Range); unit: errors
Groups:
- Placebo: Children participated in a double blind placebo controlled crossover study comparing one week of treatment with the optimal dose of OROS methylphenidate with one week of treatment with placebo. The order of administering OROS-methylphenidate versus placebo was randomized and counterbalanced across participants. At the end of each week the child's performance on different domains of attention and executive functioning was assessed.
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 29 | 29
errors
  Omission Errors | 2 [0 to 31] | 4.5 [0 to 42]
  Commission Errors | 3 [1 to 143] | 10.5 [0 to 164]
Statistical Analysis 1: Comparison: Medication vs Placebo; Same as described for TEA-Ch Walk, Don't Walk; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney) — Same as described for TEA-Ch Walk, Don't Walk

3. Primary Outcome: Wechsler Intelligence Scale for Children-IV, Digit Span Subtest
Description: The verbal assessment of working memory uses the digit span reversed component of the Digit Span subtest of the Wechsler Intelligence Scale for Children-IV edition (WISC-IV).Scores could range from 0 to 16 with higher scores indicating better performance.
Time Frame: 2 weeks
Population: The 30 subjects who completed both arms of the crossover analysis
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 5.5 [0 to 10] | 5.0 [3 to 9]
Statistical Analysis 1: Comparison: Medication vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — This p value is not adjusted for multiple comparisons

4. Secondary Outcome: Behavior Rating Inventory of Executive Function
Time Frame: 2 Weeks
Population: Although this was included in the protocol we have not analyzed the results of this rating scale
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: ADHD Rating Scale-IV, Parent and Teacher Version
Description: This is the parent and teacher version of the ADHD Rating Scale-IV. The scale has 2 subscales, one for inattention and one for hyperactivity-impulsivity. The scores provided are percentile scores and can range from 1 to 99 percent. Higher scores indicate more problems in inattention or with hyperactivity-impulsivity
Time Frame: 2 Weeks
Population: We had complete data for all 30 subjects for the parent rating scale. We only had 24 sets of complete data for the teacher rating scale as some teachers did not return a rating scale when the subject was on both medication and placebo
Measure: Mean (Standard Deviation); unit: Percentile
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 30 | 30
Percentile
  Parent Inattention Rating | 70.6 (23.9) | 92.6 (9.0)
  Parent Hyperactivity-Impulsivity Rating | 64.8 (26.5) | 89.6 (13.1)
  Teacher Inattention Rating | 61.1 (23.2) | 73.3 (19.9)
  Teacher Hyperactivity-Impulsivity Rating | 58.1 (22.1) | 75.2 (19.8)
Statistical Analysis 1: Comparison: Medication vs Placebo; A paired t-test was used to compare the medication versus placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — We did not correct for multiple comparisons; We used a paired t-test

6. Other Pre Specified Outcome: Stimulant Side Effect Rating Scale
Description: Parents rate 16 possible stimulant side effects on a 10 point likert scale from 0-9 with 0 indicating no side effects and 9 indicating more severe symptoms.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 28 | 28
Units on a scale
  Insomnia | 2.8 (2.3) | 1.2 (2.1)
  Nightmares | 0.3 (0.9) | 0.2 (0.8)
  Stares/Day Dreams | 1.1 (1.7) | 0.8 (1.3)
  Talks less with others | 1 (1.7) | 0.4 (0.8)
  Uninterested in others | 0.8 (1.4) | 0.3 (0.7)
  Decreased appetite | 3.4 (2.7) | 1 (1.8)
  Irritable | 2.6 (2.4) | 1.7 (1.9)
  Stomachaches | 1.5 (2.5) | 0.5 (1.2)
  Headaches | 0.9 (1.8) | 0.3 (0.9)
  Drowsiness | 0.9 (2.1) | 0.3 (0.9)
  Sad | 1.6 (2) | 1 (1.8)
  Prone to Crying | 2.2 (2.8) | 1.4 (2.1)
  Anxiety | 2.3 (2.4) | 1.8 (1.9)
  Bites fingernails | 1.3 (2.4) | 0.5 (0.9)
  Euphoric | 0.5 (1.4) | 0.3 (0.7)
  Dizziness | 0.1 (0.3) | 0.04 (0.19)

7. Primary Outcome: Test of Everyday Attention for Children-Sky Search Dual Task
Description: The TEA-Ch is a battery of nine subtests designed to assess multiple attentional capacities in children 6-16y.o. The Sky Search Dual Task is a measure of sustained attention. Lower scores indicate better performance. There is not a finite range for this test and very high scores can be negative numbers.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 3.8 [-3.3 to 429] | 3.9 [-0.3 to 101]
Statistical Analysis 1: Comparison: Medication vs Placebo; Same as described for TEA-Ch: Walk, Don't Walk; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney) — Same as described for TEA-Ch: Walk, Don't Walk

8. Primary Outcome: Test of Everyday Attention for Children: Score Dual Task (DT)
Description: The TEA-Ch is a battery of nine subtests designed to assess multiple attentional capacities in children 6-16y.o. The Score DT subtest is a measure of sustained attention. and response inhibition. Scores on this subtest can range from 0 to 20 with higher scores representing better performance.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 14 [5 to 20] | 13 [3 to 19]
Statistical Analysis 1: Comparison: Medication vs Placebo; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney) — The p value adjusts for multiple comparisons

9. Primary Outcome: Test of Everyday Attention for Children: Creature Counting
Description: The TEA-Ch is a battery of nine subtests designed to assess multiple attentional capacities in children 6-16y.o. The Creature Counting subtest is a measure of attentional control. There is not a finite range for this test, but lower scores indicate better performance.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 4.9 [3.1 to 12.8] | 4.8 [3.1 to 28.2]
Statistical Analysis 1: Comparison: Medication vs Placebo; Same as described for TEA-Ch: Walk, Don't Walk; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney) — Same as described for TEA-Ch: Walk, Don't Walk

10. Primary Outcome: Test of Everyday Attention for Children: Map Mission
Description: The TEA-Ch is a battery of nine subtests designed to assess multiple attentional capacities in children 6-16y.o. The Map Mission subtest is a measure of selective attention and indicates the number of targets found in one minute. Scores on this subtest can range from 0 to over 70 with higher scores representing improved performance.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 27.5 [15 to 57] | 27 [10 to 52]
Statistical Analysis 1: Comparison: Medication vs Placebo; Same as described for TEA-Ch: Walk, Don't Walk; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney) — Same as described for TEA-Ch: Walk, Don't Walk

11. Primary Outcome: Test of Everyday Attention for Children: Sky Search
Description: The TEA-Ch is a battery of nine subtests designed to assess multiple attentional capacities in children 6-16y.o. The Sky Search subtest is a measure of selective attention. There is not a finite range of scores on this subtest, but lower scores indicate better performance.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 5.8 [2.5 to 25.4] | 4.5 [2.3 to 26]
Statistical Analysis 1: Comparison: Medication vs Placebo; Same as described for TEA-Ch: Walk, Don't Walk; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney) — Same as described for TEA-Ch: Walk, Don't Walk

12. Primary Outcome: Test of Everyday Attention for Children: Opposite Worlds
Description: The TEA-Ch is a battery of subtests designed to assess multiple attentional capacities in children 6-16y.o. The Opposite Worlds subtest is a measure of attentional control and response inhibition. There is not a finite range of scores on this test. Lower scores indicate better performance..
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Medication | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 38.5 [28 to 66] | 47.5 [27 to 63]
Statistical Analysis 1: Comparison: Medication vs Placebo; Same as described for TEA-Ch: Walk, Don't Walk; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney) — Same as described for TEA-Ch: Walk, Don't Walk

ADVERSE EVENTS:
Groups:
- OROS Methylphenidate; Placebo: Children participated in a double blind placebo controlled crossover study comparing one week of treatment with the optimal dose of OROS methylphenidate with one week of treatment with placebo. The order of administering OROS-methylphenidate versus placebo was randomized and counterbalanced across participants. At the end of each week the parents rated medication side effects on the Stimulant Side Effect Rating Scale (described previously). Score of 7-9 on this scale were considered adverse effects.
Arm/Group | OROS Methylphenidate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 20/31 | 5/31
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | OROS Methylphenidate (N=31) | Placebo (N=31)
decrease appetite (Gastrointestinal disorders) | 4/28 | 1/28 — Score of 7-9 on rating scale
Irritable (Nervous system disorders) | 3/28 | 1/28 — 7-9 on rating scale
stomachaches (Nervous system disorders) | 2/28 | 0/28 — 7-9 on rating scale
Headaches (Nervous system disorders) | 1/28 | 0/28 — 7-9 on rating scale
prone to crying (Nervous system disorders) | 4/28 | 1/28 — 7-9 on rating scale
Bites Fingernails (Psychiatric disorders) | 3/28 | 0/28 — 7-9 on rating scale
Tics/Nervous movements (Nervous system disorders) | 1/28 | 0/28 — 7-9 on rating scale
Insomnia (Nervous system disorders) | 2/28 | 2/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No